CLINICAL TRIAL: NCT05546060
Title: Efficacy and Safety of Venetoclax Combined With Dexamethasone and Etoposide in the Treatment of Hemophagocytic Lymphohistiocytosis
Brief Title: Efficacy and Safety of Venetoclax Combined With Dexamethasone and Etoposide in HLH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Professor and Head of hematology, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH20220425006/BFHHZS20220026
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic Lymphohistiocytosis; Venetoclax
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — venetoclax; Dexamethasone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax Combined With Dexamethasone and Etoposide (Experimental): Patients who met the inclusion criteria will receive venetoclax combined with dexamethasone and etoposide for 8 weeks.
  Interventions: Drug: Venetoclax; Drug: Dexamethasone; Drug: Etoposide

INTERVENTIONS:
Drug: Venetoclax — Venetoclax 100mg qd d1，200mg qd d2，400mg qd d3-56
Drug: Dexamethasone — Dexamethasone 10mg/m2 qd d1-14, 5mg/m2 qd d15-28, 2.5 mg/m2 qd d29-42, and 1.25mg/m2 qd43-56
Drug: Etoposide — Etoposide 75mg/m2 qw d1-56

SUMMARY:
This study aimed to investigate the efficacy and safety of venetoclax combined with dexamethasone and etoposide as a salvage therapy for hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
Hemophagocytic lymphohistiocytosis (HLH) is a rare and aggressive disease with high mortality and poor prognosis. The HLH-94 and HLH-04 regimens are most commonly used, but approximately 30% of the patients remain unresponsive. Currently, there is no unified evidence-based salvage treatment. There is no unified salvage regimen. This study plans to enroll 20 patients with refractory and recurrent hemophagocytic lymphohistiocytosis. Subjects will receive venetoclax combined with dexamethasone and etoposide for 8 weeks.The safety was evaluated once a week, and the efficacy was evaluated once every 2 weeks. Overall response rate will be evaluated at 8 weeks. Patients were followed up every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old, expected survival time more than 3 months;
* met HLH-2004 diagnostic criteria；
* ECOG score 0-2；
* ECG QTcF interval: male ≤450ms, female ≤470ms;
* AST and ALT ≤3.0 ULN, TB ≤1.5×ULN；serum creatinine≤1.5×ULN，or CrCL ≥ 50mL/min；INR、APTT、PT ≤1.5×ULN；
* without pregnancy or lactation, and agree to contraception during and for at least 6 months after the study；
* signed informed consent.

Exclusion Criteria:

* patients with malignancies unrelated to HLH, except for fully recovered non-melanoma skin cancer and carcinoma in situ;
* patients participated in other clinical trials within 4 weeks；
* previously treated with Bcl-2 inhibitors；
* unable to take oral medication；
* history of substance abuse or patients with mental illness；
* severe infection；
* cardiovascular disease，NYHA II-IV；
* allergic to venetoclax or etoposide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The percentage of cases with complete response (CR) and partial response (PR) after treatment in the total evaluable cases
Incidence and severity of adverse effects | 1 years
  The percentage of cases with adverse effects and its severity.

SECONDARY OUTCOMES:
Overall survival | 1 years
  OS is defined as the time from the initiaion of treatment to death from any cause or July 2025.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No